CLINICAL TRIAL: NCT04243915
Title: Effectiveness of Percutaneous Neuromuscular Electrical Stimulation on Lumbar Multifidus in Combination With a Protocol of Motor Control Exercises in Patients With Chronic Low Back Pain
Brief Title: Percutaneous Neuromuscular Electrical Stimulation in Patients With Chronic Low Back Pain
Acronym: PNMESlowback
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Josue Fernandez Carnero, PhD, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EC 01/2019
Record Dates: First submitted 2020-01-15; First posted 2020-01-28 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Low Back Pain
Keywords: Percutaneous neuromuscular electrical stimulation; Percutaneous electrical nerve stimulation; Percutaneous electrical stimulation; Motor control exercise; Multifidus; Abdominal transverse; Non-specific chronic low back pain; Transcutaneous electric nerve stimulation; Exercise therapy
MeSH Terms: conditions — Low Back Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo controlled clinical trial.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PNMES plus exercise (Experimental): 6-week intervention program with 3 treatment sessions of PNMES and motor control exercise program.
  Interventions: Other: Percutaneous neuromuscular electrical stimulation (PNMES) plus motor control exercise program
- Sham PNMES (introducing the needle) plus exercise (Sham Comparator): Sham PNMES (introducing the needle) plus motor control exercise program
  Interventions: Other: Sham PNMES (introducing the needle) plus motor control exercise program
- TENS plus exercise (Active Comparator): 6-week intervention program with 3 treatment sessions of TENS plus motor control exercise program.
  Interventions: Other: TENS plus motor control exercise program
- Placebo PNMES (without inserting the needle) plus exercise (Placebo Comparator): 6-week intervention program with 3 treatment sessions of placebo PNMES (without inserting the needle) and exercise
  Interventions: Other: Sham PNMES (without inserting the needle) plus motor control exercise program

INTERVENTIONS:
Other: Percutaneous neuromuscular electrical stimulation (PNMES) plus motor control exercise program — The technique consists of a muscular stimulation of the deep lumbar multifidus by means of a TENS current applied through four dry needling or acupuncture needles introduced by ultrasound guidance in said muscle 30 minutes. This will add to a protocol of motor control exercises for deep abdominal and lumbar muscles.
  Other Names: Percutaneous electric nerve stimulation (PENS)
  Arms: PNMES plus exercise
Other: Sham PNMES (introducing the needle) plus motor control exercise program — The same procedure will be performed as in the experimental treatment, but in this case, the electric current will be placebo and only the first 15 seconds will slightly notice it. This will add to a protocol of motor control exercises for deep abdominal and lumbar muscles.
  Other Names: Sham PENS
  Arms: Sham PNMES (introducing the needle) plus exercise
Other: TENS plus motor control exercise program — Transcutaneous electrical nerve stimulation will be applied through 4 patches / adhesives placed in your lower back for 30 minutes. This will add to a protocol of motor control exercises for deep abdominal and lumbar muscles.
  Other Names: TENS
  Arms: TENS plus exercise
Other: Sham PNMES (without inserting the needle) plus motor control exercise program — The same procedure will be performed as in the experimental treatment, but in this case, the needle will not be inserted and the electric current will be placebo and only the first 15 seconds will slightly notice it. This will add to a protocol of motor control exercises for deep abdominal and lumbar muscles.
  Other Names: Sham PENS
  Arms: Placebo PNMES (without inserting the needle) plus exercise

SUMMARY:
Chronic low back pain is a common musculoskeletal condition affects the general population. Low back pain constitutes a major burden to health care system and society. Several authors have found that the deep abdominal muscles and multifidus are affected in low back pain. Dry needling has shown improve the cross-sectional area of the multifidus. Percutaneous electrical nerve stimulation has shown reduce pain in several conditions. There are not studies that had investigated the impact of percutaneous neuromuscular electrical stimulation (PNMES) in the deep muscles in patients with chronic low back pain.

Hypothesis: PNMES in the multifidus muscle plus motor control exercise program in patients with chronic low back pain is better than sham PNMES plus exercise and transcutaneous electrical nerve stimulation (TENS) plus exercise

DETAILED DESCRIPTION:
Randomized, double-blind, placebo controlled clinical trial, using percutaneous neuromuscular electrical stimulation (PNMES). PNMES is technique to provide a transcutaneous electrical nerve stimulation current throughout needling filaments place close to the nerve.

Study Aims:

Aim #1: The primary aim of the study is to compare the effect of the short, medium and long-term of PNMES on muscle activation (increased cross-sectional area in activation) and the function of multifidus and abdominal transverse muscle in patients with chronic low back pain with random assignment to four treatments: PENS plus motor control exercise program or Sham PNMES (introducing the needle) plus motor control exercise program or Transcutaneous Electrical Nerve Stimulation (TENS) plus motor control exercise program or Sham PNMES (without inserting the needle) plus motor control exercise program.

Aim #2: The secondary aim of the study is to compare the effect of the short, medium and long-term of PNMES on pain as measured by visual analogue scale (VAS), chronic Pain Grade Questionnaire, pressure pain threshold (PPT), area and distribution of pain, conditioned pain modulation and temporal summation in patients with chronic low back pain with random assignment to four treatments: PNMES plus motor control exercise program or Sham PNMES (introducing the needle) plus motor control exercise program or Transcutaneous Electrical Nerve Stimulation (TENS) plus motor control exercise program or Sham PNMES (without inserting the needle) plus motor control exercise program.

Aim #3: To compare the effect of the short, medium and long-term of PNMES on disability as measured by Oswestry Disability Index, strength and quality of life with random assignment to four treatments: PENS plus motor control exercise program or Sham PNMES (introducing the needle) plus motor control exercise program or Transcutaneous Electrical Nerve Stimulation (TENS) plus motor control exercise program or Sham PNMES (without inserting the needle) plus motor control exercise program.

Aim #4: To estimate the immediate effects of the PNMES technique after the first session.

Aim #5: To determine if psychological factors (anxiety, depression, kinesiophobia and catastrophism) change with any of the treatments and if is related with the primary and secondary outcomes.

Aim #6: To evaluate the change perceived by the patient measured with Global Rating of Change Scale (GROC).

Aim Aim #7: Validation of placebo groups by assessing patient blindness

ELIGIBILITY:
Inclusion Criteria:

- Low back pain more than 90 days of evolution

Exclusion Criteria:

* Spondylarthrosis
* History of fractures, luxations, surgery and/or musculoskeletal disorders in low back and lower limb.
* Leg pain or neuropathic pain (LANSS <12).
* Neurological disorders, inflammatory and/or degenerative diseases.
* Having received as treatment techniques that involve needles on the previous 6 months to study enrollment or having received percutaneous electrical stimulation as a treatment before.
* Physiotherapy treatment in the last 4 weeks.
* Specific lumbar pathology, fibromyalgia, unstable cardiovascular diseases, pregnant women or under suspect of pregnancy.
* Contraindications of needle's insertions: anticoagulant therapy, needle phobia, diabetes, hypothyroidism, lymphoedema, muscular diseases).
* Contraindications of electrical current.
* Drugs: morphine or opioids drugs.
* Depression
* Judicial dispute

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2021-04-10 (Actual); Primary Completion 2024-06-10 (Estimated); Study Completion 2024-12-10 (Estimated)

PRIMARY OUTCOMES:
Increased cross-sectional area in activation | Baseline, one hour from baseline after PNMES treatment 1, 6 weeks from baseline, 18 weeks from baseline and 30 weeks from baseline
  The increase in height from the resting position to the submaximal contraction in the lumbar multifidus will be measured
Changes in the measurements of the multifidus and tranverse of the abdomen at rest. | Baseline, one hour from baseline after PNMES treatment 1, 6 weeks from baseline, 18 weeks from baseline and 30 weeks from baseline
  Changes in the height of the multifidus at rest

SECONDARY OUTCOMES:
Intensity of Pain | (Baseline, one hour from baseline after PNMES treatment 1 (only at rest), 6 weeks from baseline, 18 weeks from baseline and 30 weeks from baseline
  Will be measure with a line of 100 mmm (0 - no pain to 100- the worst pain) at rest and his best and worst pain in the last 24 hours.
Pressure pain threshold using an algometer | Baseline, one hour from baseline after PNMES treatment 1, 6 weeks from baseline, 18 weeks from baseline and 30 weeks from baseline
  Measurement of pressure pain threshold in the paravertebral muscles, in the spinous process of L4, and the tibialis anterior muscle.
Temporal summation | Baseline, one hour from baseline after PNMES treatment 1, 6 weeks from baseline, 18 weeks from baseline and 30 weeks from baseline
  Ten consecutives pressure pain stimulus will be conducted, pain intensity in the first, fifth and tenth will be asked. The difference from 1 to 10 will be the value that reports on the state of excitability of the posterior horn of the medulla
Conditioned pain modulation | Baseline, one hour from baseline after PNMES treatment 1, 6 weeks from baseline, 18 weeks from baseline and 30 weeks from baseline
  First, pressure pain stimulus (test stimulus) will be conducted in the distal phalanx of the thumb. Second, occlusion cuff will be inflated around the arm of patient until the patient feeling a painful intensity (conditioned stimulus) of 6/10. Finally, after 30 seconds the stimulus will be done. The difference in the mean value of the initial algometry with the mean value of algometry during the conditioning stimulus will indicate the state of the descending pain inhibitory system.
Pain Grade Questionnaire | Baseline, 6 weeks from baseline, 18 weeks from baseline and 30 weeks from baseline
  The scale assesses two dimensions: the intensity of pain and pain related to disability. It can be used in any chronic pathology including musculoskeletal problems and low back pain. It allows the graduation of the severity of chronic pain and the subsequent analysis of the qualitative changes for that pain. The scale has 7 items, which are of the Likert type of 11 points, with a total range of 0 to 70 points.
Oswestry Disability Index or Oswestry Low Back Pain Disability Questionnaire | Baseline, 6 weeks from baseline, 18 weeks from baseline and 30 weeks from baseline
  The Oswestry Disability Index (ODI) is a validated, self-reported instrument used by clinicians and researchers to quantify disability for low back pain.
  The self-completed questionnaire contains ten topics concerning intensity of pain, lifting, ability to care for oneself, ability to walk, ability to sit, sexual function, ability to stand, social life, sleep quality, and ability to travel. Each topic category is followed by 6 statements describing different potential scenarios in the patient's life relating to the topic. The patient then checks the statement which most closely resembles their situation. Each question is scored on a scale of 0-5 with the first statement being zero and indicating the least amount of disability and the last statement is scored 5 indicating most severe disability. The scores for all questions answered are summed, then multiplied by two to obtain the index (range 0 to 100). Zero is equated with no disability and 100 is the maximum disability possible.
Short form 12 (SF-12) health survey (health-related quality of life) | Baseline, 6 weeks from baseline, 18 weeks from baseline and 30 weeks from baseline
  The SF-12 is a validated, health-related quality-of-life questionnaire consisting of twelve questions that measure eight health domains to assess physical and mental health. Physical health-related domains include General Health (GH), Physical Functioning (PF), Role Physical (RP), and Body Pain (BP). Mental health-related scales include Vitality (VT), Social Functioning (SF), Role Emotional (RE), and Mental Health (MH). The instrument has been validated across a number of chronic diseases and conditions. The response options of the SF-12 v2 form Likert-type scales that evaluate intensity or frequency. The number of answer options ranges from three to six, depending on the item, and each question is given a value which is then transformed into a scale from 0 to 100.
Kinesiophobia | Baseline, 6 weeks from baseline, 18 weeks from baseline and 30 weeks from baseline
  Tampa Scale for Kinesiophobia. To assess the fear of movement and pain-related fear. The 11 items are scored 1-4, with total scores ranging from 11 to 44. The addition of all the points obtained from each of the items results in the level of kinesiophobia, with higher scores indicating greater perceived kinesiophobia
Pain catastrophizing | Baseline, 6 weeks from baseline, 18 weeks from baseline and 30 weeks from baseline
  Pain Catastrophizing Scale (PCS). This tool is a 13-item questionnaire designed to measure the three components of pain-related catastrophizing: rumination, magnification, and helplessness, resulting in a unique score. Each item is responded to on a 5-point scale (0 not at all, 4 all the time) relating the degree to which the individual experiences a thought or feeling of a painful situation.
The Becks Depression Inventory-II | Baseline, 6 weeks from baseline, 18 weeks from baseline and 30 weeks from baseline
  The Becks Depression Inventory-II is a validated, self-administered questionnaire consisting of 21 multiple choice questions. It is one of the most commonly used instruments to measure the severity of a depression. Possible scores range from 0 (no depression) to 63 (severe depression).
Anxiety | Baseline, 6 weeks from baseline, 18 weeks from baseline and 30 weeks from baseline
  The state-trait anxiety inventory (STAI) is a questionnaire that measures trait anxiety (a personality factor that predisposes the patient to suffer from anxiety) and the state of anxiety (environmental factors that protect or generate anxiety). Each of the two sub-scales (trait anxiety and state anxiety) consists of 20 items, ranging from 0 (nothing) to 3 (a lot).
Global Rating of Change Scale | Baseline, 6 weeks from baseline, 18 weeks from baseline and 30 weeks from baseline
  Global Rating of Change (GRoC) scales provide a means of measuring self-perceived change in health status. Possible scores range from -5 (very much worse), through 0 (unchanged) to +5 (completely recovered).
Blinding the patient | 1 hour from baseline after the PNMES treatment 1, 2 weeks from baseline after the second PNMES treatment and 4 weeks from baseline after the third PNMES treatment
  The patients of the sham groups will be asked after the interventions of PNMES if they belonged to the group of deep electro-stimulation, being able to content: Sure that yes, moderately that yes, I do not know, moderately that no or sure that no.
Central Sensitization Inventory | Baseline, 6 weeks from baseline, 18 weeks from baseline and 30 weeks from baseline
  The Spanish version of the Central Sensitisation Inventory will be used to identify symptoms related to central sensitisation. It is a self-report questionnaire that assesses a total of 25 sensitisation-associated symptoms on a 5-point Likert scale. The total score ranges from 0 to 100, where >40/100 points suggest the presence of sensitisation-associated symptoms. It has been found to have high reliability and validity.

CONTACTS AND LOCATIONS:
Overall Officials: Josue Fernández-Carnero, PhD, Principal Investigator — Universidad Rey Juan Carlos
Locations (1):
- Universidad Rey Juan Carlos, Alcorcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No